CLINICAL TRIAL: NCT00940355
Title: Secondary Prevention of Problems in Health Status in Patients With COPD by Early Detection, Motivational Intervention to Engage in Treatment by the Patient, and by Individualized Treatment
Brief Title: Secondary Prevention of Problems in Health Status in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: PICASSO: Partners in Care Solutions for COPD (Other)
Responsible Party: Dr. J.H.M.M. Vercoulen, Radboud University Nijmegen Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PICASSO 06-009; NTR1844
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Health Status
Keywords: COPD; Health Status; Intervention; Secondary prevention; patient-tailored treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention pulmonary nurse (Experimental): group III: intervention conducted by a pulmonary nurse, directed at increasing awareness of problems in health status, increasing motivation to engage in additional treatment, and improving health status.
  Interventions: Behavioral: Intervention pulmonary nurse
- Usual care (No Intervention): group II: usual care as delivered by the outpatient clinic.

INTERVENTIONS:
Behavioral: Intervention pulmonary nurse — The intervention is conducted by a pulmonary nurse, directed at increasing awareness of problems in health status, and increasing motivation to engage in additional treatment, and improving health status.
  Arms: Intervention pulmonary nurse

SUMMARY:
The purpose of this study is to determine the effectiveness of an intervention conducted by a pulmonary nurse in patients with COPD.

The hypothesis is that in a sample of COPD patients with clinically relevant problems in health status (physiological functioning, symptoms, functional impairment and quality of life), a motivational intervention conducted by a pulmonary nurse will lead to patient-tailored treatment and an improved health status.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a disease state characterized by airflow that is not fully reversible. Besides problems in physiological functioning, the patient also can experience symptoms, functional impairment and a diminished quality of life (see Vercoulen et al., 2008). Problems in the three latter domains of health status are hardly recognized in usual care, and remain untreated until escalated. This is mainly caused by two phenomena: doctor delay and patient delay. Doctor delay: the physician does not directly identify symptoms, functional impairment, and problems in quality of life. Patient delay: the patient does not report problems in these health status domains.

What is necessary is a screening instrument that can be used in routine care and identifies patients with problems in the four domains of health status. If clinically relevant problems exists, and additional treatment is recommended, an intervention by the pulmonary nurse is indicated. This intervention is directed at increasing awareness of existing problems and motivating the patient for additional treatment. By means of the screening and intervention, problems in health status are detected and treated early, before escalation. Treatment is patient-tailored, based on the existing problems in the four domains of health status, eventually leading to an improved health status.

A randomized controlled trial is conducted to test the hypothesis described above. Based on the independent clinical interpretation of the PatientProfileChart (see Peters et al., 2009) by three professionals, patients are assigned to one of the following groups: 1. Patients with no clinically relevant problems in health status (group I), and 2. Patients with clinically relevant problems in health status (group II/III). Patients with clinically relevant problems in health status are randomized to a control group (group II: usual care as delivered by the outpatient clinic) and the experimental group (group III: intervention conducted by a pulmonary nurse, directed at increasing awareness of problems in health status, increasing motivation to engage in additional treatment, and improving health status).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Written informed consent

Exclusion Criteria:

* Not able to adhere to study protocol
* Not competent enough in understanding Dutch language
* Participation in pulmonary rehabilitation program within previous 6 months
* Current participation in other research study in COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Physiological Functioning: TLC% predicted, RV% predicted, FEV1% predicted, BMI | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
Symptoms: Physical Activity Rating Scale Dyspnoea- Global Dyspnoea Activity and Global Dyspnoea Burden, Dyspnoea Emotions Questionnaire - Frustration and Anxiety, Checklist Individual Strength - Fatigue | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
Quality of Life: Beck Depression Inventory Primary Care, Satisfaction with Life Scale, Satisfaction Physical, Satisfaction Future, Satisfaction Spouse and Satisfaction Social | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
Functional Impairment: Quality of Life for Respiratory Illness Questionnaire - General Activities, Sickness Impact Profile - Home Management and Ambulation | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
The number of additional treatments | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III

SECONDARY OUTCOMES:
Smoking status | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
Patient satisfaction with treatment | T1 (after 6 months) T2 (after 12 months). T1: group II/III T2 group I/II/III
Sociodemographic variables (i.e. sex, age, education, personal situation, work situation) | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
Clinical variables (i.e. comorbidity, previous and current treatments, hospitalization) | T0 (baseline), T1 (after 6 months) T2 (after 12 months). T0: group I/II/III T1: group II/III T2 group I/II/III
Accuracy of diagnostic properties of the PatientProfileChart | T0 (baseline), T0: group I/II/III

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Daudey, MSc., Principal Investigator — Radboud University Nijmegen Medical Center, department of Medical Psychology & department of Pulmonary Diseases; Jan Vercoulen, Dr., Study Director — Radboud University Nijmegen Medical Center, department of Medical Psychology & department of Pulmonary Diseases; Jan Vercoulen, Dr., Study Chair — Radboud University NIjmegen Medical Center, Department of Medical Psychology & department of Pulmonary Diseases
Locations (1):
- Radboud University Nijmegen Medical Center, department of Pulmonary Diseases, Groesbeek, Netherlands

REFERENCES:
- [Background] Vercoulen JH, Daudey L, Molema J, Vos PJ, Peters JB, Top M, Folgering H. An Integral assessment framework of health status in chronic obstructive pulmonary disease (COPD). Int J Behav Med. 2008;15(4):263-79. doi: 10.1080/10705500802365474. PMID 19005926
- [Background] Peters JB, Daudey L, Heijdra YF, Molema J, Dekhuijzen PN, Vercoulen JH. Development of a battery of instruments for detailed measurement of health status in patients with COPD in routine care: the Nijmegen Clinical Screening Instrument. Qual Life Res. 2009 Sep;18(7):901-12. doi: 10.1007/s11136-009-9502-2. Epub 2009 Jun 19. PMID 19543807